CLINICAL TRIAL: NCT01510301
Title: Mastery and Autonomy in Management of Hypertension With a Mobile Self-report System
Brief Title: Mobile Phone in Hypertension Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MIHM
Record Dates: First submitted 2012-01-11; First posted 2012-01-16 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Hypertension
Keywords: Self-report; Self-management; Hypertension; Adherence; Cell phone; Drug treatment; Medical Adherence
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Self-report (Other)
  Interventions: Device: Mobile phone-based self-report system, electronic Patient-Reported Outcomes Measure (e-PROM)

INTERVENTIONS:
Device: Mobile phone-based self-report system, electronic Patient-Reported Outcomes Measure (e-PROM) — To test an electronic Patient-Reported Outcomes Measure (e-PROM) intended to assess patients' daily perceptions of symptoms and wellbeing, as well as self-measured blood pressure, treatment side-effects and medicine intake;
  * Explore patient interactions (learning and understanding) with an internet-reporting system providing structured feedback of e-PROM results to examine if such feedback is useful in improving adherence;
  * Explore patient-physician/nurse interactions to examine if structured feedback of e-PROM results serves as a useful complement to support consultations regarding treatment monitoring and adherence.

SUMMARY:
The purpose of this study is to examine if a mobile phone-based self-report system, using the patient's own mobile phone, will improve adherence to treatment of hypertension and lead to personal involvement of the patient in the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of arterial hypertension
* Prescribed antihypertensive treatment
* Alert and oriented
* Swedish-speaking
* Access to a functioning cell phone
* Agreeing to regular controls at the National Prescribed Drug Register of drugs

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Adherence to antihypertensive medication | 8 weeks
  Adherence to antihypertensive medication will be checked through a question in the cell phone and evaluation of patient´s use of antihypertensive medication will be checked from the National Prescribed Drug Register of drugs. Twenty patient-physician/nurse consultations will be audio/video-recorded at regularly scheduled appointments to obtain authentic evidence of the use of the self-reports in clinical practice. The outcomes will include blood pressure measurement, registration of self-reported symptoms and discourse analyses.

SECONDARY OUTCOMES:
Systolic blood pressure | 8 weeks
  Change in systolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Karin I Kjellgren, professor, Principal Investigator — Göteborg University
Locations (1):
- University of Gothenburg, Gothenburg, Box 457, Sweden

REFERENCES:
- [Result] Bengtsson U, Kasperowski D, Ring L, Kjellgren K. Developing an interactive mobile phone self-report system for self-management of hypertension. Part 1: patient and professional perspectives. Blood Press. 2014 Oct;23(5):288-95. doi: 10.3109/08037051.2014.883203. Epub 2014 Feb 24. PMID 24564289
- [Result] Bengtsson U, Kjellgren K, Hofer S, Taft C, Ring L. Developing an interactive mobile phone self-report system for self-management of hypertension. Part 2: content validity and usability. Blood Press. 2014 Oct;23(5):296-306. doi: 10.3109/08037051.2014.901009. Epub 2014 May 1. PMID 24786778
- [Result] Hallberg I, Taft C, Ranerup A, Bengtsson U, Hoffmann M, Hofer S, Kasperowski D, Makitalo A, Lundin M, Ring L, Rosenqvist U, Kjellgren K. Phases in development of an interactive mobile phone-based system to support self-management of hypertension. Integr Blood Press Control. 2014 May 7;7:19-28. doi: 10.2147/IBPC.S59030. eCollection 2014. PMID 24910510
- [Result] Hallberg I, Ranerup A, Kjellgren K. Supporting the self-management of hypertension: Patients' experiences of using a mobile phone-based system. J Hum Hypertens. 2016 Feb;30(2):141-6. doi: 10.1038/jhh.2015.37. Epub 2015 Apr 23. PMID 25903164
- [Result] Bengtsson U, Kjellgren K, Hallberg I, Lindwall M, Taft C. Improved Blood Pressure Control Using an Interactive Mobile Phone Support System. J Clin Hypertens (Greenwich). 2016 Feb;18(2):101-8. doi: 10.1111/jch.12682. Epub 2015 Oct 12. PMID 26456490
- [Result] Ruiz-Hurtado G, Ruilope LM. New Strategy to Control Blood Pressure: Interactive Mobile Phone Support. J Clin Hypertens (Greenwich). 2016 Feb;18(2):109-10. doi: 10.1111/jch.12683. Epub 2015 Oct 14. No abstract available. PMID 26462732
- [Derived] Taft C, Hallberg I, Bengtsson U, Manhem K, Kjellgren K. Links between blood pressure and medication intake, well-being, stress, physical activity and symptoms reported via a mobile phone-based self-management support system: a cohort study in primary care. BMJ Open. 2018 Aug 23;8(8):e020849. doi: 10.1136/bmjopen-2017-020849. PMID 30139897
- [Derived] Bengtsson U, Kjellgren K, Hallberg I, Lundin M, Makitalo A. Patient contributions during primary care consultations for hypertension after self-reporting via a mobile phone self-management support system. Scand J Prim Health Care. 2018 Mar;36(1):70-79. doi: 10.1080/02813432.2018.1426144. Epub 2018 Jan 18. PMID 29343156